CLINICAL TRIAL: NCT02954679
Title: French Study on COgnitive Enhancement and Consumption of Psychoactive Substances Among Youth Students (Enquête Nationale Sur le Dopage Intellectuel et Les Consommations de Substances Psychoactives Chez Les Jeunes étudiants)
Brief Title: French Study on COgnitive Enhancement and Consumption of Psychoactive Substances Among Youth Students
Acronym: ENQUETE-COSYS
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Mission Interministérielle de Lutte contre les Drogues et les Conduites Addictives - MILDECA (Unknown); Agence Nationale de sécurité du Médicament (Other)
Responsible Party: Sponsor
Other Study IDs: UC1602
Record Dates: First submitted 2016-11-02; First posted 2016-11-03 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2017-04

CONDITIONS: Psychoactive Substances Consumption; Substance-related Disorder; Off Label-use; Cognitive Enhancement
Keywords: Psychoactive Substances Consumption; Substance-related Disorder; Off label-use; Cognitive Enhancement; Students; Doping; Stimulants; Drug abuse; Methylphenidate; Addictovigilance; CEIP
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Online self-administrated and anonymous survey questionnaire — The study will be conducted during a period of 3 years, between September 2016 and September 2019, according to a standardized methodology identical in every school involved and a procedure based on an online self-administrated and anonymous survey questionnaire. The questionnaire, elaborated on Limesurvey®, will be available for two successive academic years for all students aged more than 18 years old.

SUMMARY:
This descriptive and declarative study will help to find out consumption rates, all psychoactive substances taken together, among 18-25 year olds. More specifically, it will allow assessment of the extent of the cognitive enhancement phenomenon among students in France (including study of misuse of methylphenidate (MPH) and modafinil in improvement of cognitive performance).

DETAILED DESCRIPTION:
This descriptive and declarative study will help to find out consumption rates, among 18-25 year olds, all psychoactive substances (PAS) taken together. More specifically, it will allow assessment of the extent of the cognitive enhancement phenomenon among students in France (including study of misuse of methylphenidate (MPH) and modafinil, two drugs diverted from their indications for improvement of cognitive performance).

Since Faculties of Sciences and Technics of Physical and Sports Activities (UFR STAPS) are involved in the study, the issue of doping in Sports will also be addressed.

The main aim of this national study will be to assess for two successive academic years the proportion and motives of consumption of PAS as part of cognitive enhancement among students in real life.

Secondary aims will be: assessing consumption of PAS and desired effects when such consumption beyond cognitive enhancement (experimental, recreational, abusive or therapeutic use) but also comparing PAS uses in terms of a variety of characteristics (sex, age, field, year of study) and finally to consider more broadly the health of students in a doping behavior (impact of the use of products on health, whether cognitive enhancement is found to be ethically acceptable or not).

The study will be conducted during a period of 3 years, between September 2016 and September 2019, according to a standardized methodology identical in every school involved and a procedure based on an online self-administrated and anonymous survey questionnaire. The questionnaire, elaborated on Limesurvey®, will be available for two successive academic years for all students aged more than 18 years old. It is set up and hosted on a secured high-capacity web server via the website of AP-HP.

The study will also search to assess the level of representation of the sample of respondents regarding the general population of students. Various criteria: the proportion of subjects by field, the proportion of respondents by study year and the sex ratio will be compared to data of general statistics from the Ministry of Research and Higher Education. A representative sample will allow us to assimilate our respondents to the general population of students and estimate the prevalence of PAS consumption among students.

METHODS

For each product, a descriptive analysis of frequency will be done (consumption pattern, consumer's opinion, feeling of dependency, efficacy of the product). For those most frequently used, complementary analysis will be done in order to identify particular profiles.

On the statistical level, univariate analysis will be performed using the Chi-square test and analysis of variance. Then, multivariate analysis will allow us to study independent factors such as age and study year for instance.

The number of respondents expected is approximately 30 000. The sample will also allow us to identify factors associated with PAS consumption (MPH or modafinil particularly) by multivariate modeling using a "split" of the sample procedure with one half used for the construction of the model and the other for its validation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged more than 18 years old
* Students (University, BTS, Grandes Ecoles, IFSI, preparatory classes) registered in the ongoing year

Exclusion Criteria:

- Minor subjects

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students 18-25 year olds in Faculties of Sciences and Technics of Physical and Sports Activities (UFR STAPS) are involved in the study, the issue of doping in Sports will also be addressed.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

PRIMARY OUTCOMES:
Rate of PAS use for the purpose of cognitive enhancement among students since the beginning of the school year, depending on the school | between January and April 2017 and January and April 2018

SECONDARY OUTCOMES:
Rate of use for each PAS | between January and April 2017 and January and April 2018
Motives of consumption : hedonic (festive, recreational, experimental, boredom management) | between January and April 2017 and January and April 2018
Motives of consumption : performance (creativity, sports, cognition) | between January and April 2017 and January and April 2018
Motives of consumption : therapeutic (sleep disorder, anxiety, sadness, weight control) | between January and April 2017 and January and April 2018
Motives of consumption : social (making friends, being noticed, assertion of identity)control) | between January and April 2017 and January and April 2018
Consumption pattern (dose, route of administration, frequency, way to obtain, associated drugs, period) | between January and April 2017 and January and April 2018
Comparison PAS uses in terms of a variety of characteristics of subjects (sex, age, sector, year of study). | between January and April 2017 and January and April 2018

CONTACTS AND LOCATIONS:
Overall Officials: DJEZZAR Samira, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Clermont-Ferrand - service de santé publique, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Batisse A, Leger S, Vicaut E, Gerbaud L, Djezzar S. COgnitive enhancement and consumption of psychoactive Substances among Youth Students (COSYS): a cross-sectional study in France. Public Health. 2021 May;194:75-78. doi: 10.1016/j.puhe.2021.02.036. Epub 2021 Apr 14. PMID 33865150